CLINICAL TRIAL: NCT01755806
Title: Comparison of Aortic Root Dimension Changes During Cardiac Cycle Between the Patients With and Without Aortic Valve Calcification Using ECG-gated 64-slice and Dual-source 256-slice Computed Tomography Scanners: Results of a Multicenter Study
Status: Completed | Type: Observational
Sponsor: Modarres Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ModarresH_001
Record Dates: First submitted 2012-12-17; First posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Aortic Valve Calcification
Keywords: Aortic annulus; Aortic calcification; Multislice computed tomography; Cardiac cycle
MeSH Terms: conditions — Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aortic root dimension change: those without aortic valve calcification
- aortic root dimension change, aortic valve calcium score: those with aortic valve calcification

SUMMARY:
This study seeks to compare aortic dimension changes during cardiac cycle in patients with and without aortic valve calcification and to evaluate its correlation with aortic valve calcium score in former group.

DETAILED DESCRIPTION:
The study population comprised 104 patients referred to three cardiac imaging centers for coronary multislice computed tomography, including 52 patients with aortic valve calcification as the study group and 52 subjects without evidence of calcification in their aortic valve, who served as a control group. Data were reconstructed at each 10% of RR-interval during the cardiac cycle and reconstructed images at 30-35% and 70-75% of R-R intervals were obtained, representing systole and diastole, respectively. For diastolic phase, in most cases images at 70% were acquired. Thereafter, acquired images were transferred to a single remote workstation for post-processing and subsequent off-line analysis.

ELIGIBILITY:
Inclusion Criteria:

- Patients referring for multislice coronary computed tomography for any reason

Exclusion Criteria:

* Arrhythmia
* Hypertrophic cardiomyopathy
* Aneurysm formation of ascending aorta
* Marfan's disease
* Ehlers-Danlos syndrome
* History of coronary artery bypass surgery
* History of coronary stenting
* Aortic valve surgery
* Thoracic aorta surgery
* Aortic valve stenosis

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referring for coronary CT angiography
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evidence of aortic root dimension change confirmed by multislice CT in systolic phase (30% of R-R interval) compared to diastolic phase (70% of R-R interval) after retrospective ECG gating | during a few heat beat (8 to 13 seconds)
  Detailed information about aortic root dimension changes during cardiac cycle has become of utmost interest especially after introduction of transcatheter aortic valve implantation (TAVI) as an alternative therapeutic procedure in patients with severe aortic stenosis, in that paravalvular regurgitation and procedural failure will ensue from errors in selecting the appropriate prosthesis size

CONTACTS AND LOCATIONS:
Locations (3):
- Iran (3):
  - Modarres Hospital, Tehran
  - Day General Hospital, Tehran
  - Rajaie Cardiovascular medical and Research Center, Tehran

REFERENCES:
- [Derived] Arjmand Shabestari A, Pourghorban R, Tehrai M, Pouraliakbar H, Faghihi Langroudi T, Bakhshandeh H, Abdi S. Comparison of aortic root dimension changes during cardiac cycle between the patients with and without aortic valve calcification using ECG-gated 64-slice and dual-source 256-slice computed tomography scanners: results of a multicenter study. Int J Cardiovasc Imaging. 2013 Aug;29(6):1391-400. doi: 10.1007/s10554-013-0217-7. Epub 2013 Apr 13. PMID 23584562